CLINICAL TRIAL: NCT02087202
Title: Hyperalgesia and NMDA Receptor Antagonist
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Kim Mihyun, clinical professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: hyperalgesia
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Pain
Keywords: pain
MeSH Terms: conditions — Pain | interventions — Magnesium Sulfate; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- magnesium (Experimental): magnesium is added perioperatively to those patients undergoing staged total knee arthroplasty and other surgeries.
  Interventions: Drug: Magnesium Sulfate
- ketamine (Experimental): ketamine is administered to those patients undergoing stated TKA and other operations.
  Interventions: Drug: ketamine
- control (Placebo Comparator): normal saline (placebo) is administered to the patients.

INTERVENTIONS:
Drug: Magnesium Sulfate — magnesium sulfate is added to the patients
  Arms: magnesium
Drug: ketamine — ketamine is added to the patients.
  Arms: ketamine

SUMMARY:
NMDA receptor is administered and postoperative remote hyperalgesia is investigated.

DETAILED DESCRIPTION:
NMDA receptor is adminstered and postoperative tertiary hyperalgesia is investigated.

QST and pain measures for remote hyperalgesia are compared between control and magnesium or ketamine group.

ELIGIBILITY:
Inclusion Criteria:

* ASA1-2

Exclusion Criteria:

* contraindication to the study drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
pain | until 1 month from the end of the operation
  pain (QST and pain measures )until 1 month from the end of the operation